CLINICAL TRIAL: NCT07306741
Title: Cognitive Versus Image Guided Fusion Transrectal Prostatic Biopsy for the Detection of Prostate Cancer
Brief Title: Cognitive and Fusion Prostatic Biopsy
Acronym: CTB-FTB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mohammed, ASSISTANT LECTURER, Menoufia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: UROL 22
Record Dates: First submitted 2025-11-27; First posted 2025-12-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Cognitive-Targeted Biopsy; Magnetic Resonance Imaging-Ultrasound Fusion Biopsy; Multiparametric Magnetic Resonance Imaging; Transrectal Prostate Biopsy; Prostate Cancer Detection; Diagnostic Accuracy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential cognitive-targeted biopsy followed by fusion-targeted biopsy (Experimental): Participants will undergo a cognitive-targeted prostate biopsy followed immediately by a fusion-targeted prostate biopsy during the same session. Each participant will receive both biopsy techniques sequentially, allowing within-subject comparison. Participants will be assigned to one of two surgeons using a blinded randomization process; however, all participants will receive the same intervention protocol.
  Interventions: Procedure: Cognitive-targeted prostate biopsy

INTERVENTIONS:
Procedure: Cognitive-targeted prostate biopsy — Participants will undergo a cognitive-targeted prostate biopsy followed immediately by a fusion-targeted prostate biopsy during the same session.
  Other Names: Fusion-targeted prostate biopsy

SUMMARY:
The goal of this study is to compare two different prostate biopsy techniques used to detect prostate cancer. These techniques are cognitive-targeted biopsy (CTB) and magnetic resonance imaging-ultrasound fusion-targeted transrectal biopsy (FTB). Both methods aim to improve the accuracy of prostate cancer detection by targeting suspicious areas identified on prostate imaging. This study will compare how accurately each technique detects prostate cancer, the pathological findings obtained from each biopsy method, and how operator performance may influence the procedure. The information gained from this study may help improve prostate cancer diagnosis and guide future biopsy practices.

DETAILED DESCRIPTION:
This study will be conducted in the urology department, Menoufia University, and will include biopsy-naïve patients with clinical suspicion of prostate cancer. Suspicion will be based on abnormal digital rectal examination (DRE) findings and prostate-specific antigen (PSA) levels between 4 and 20 nanograms per milliliter (ng/mL).

All eligible patients will undergo multiparametric magnetic resonance imaging (mpMRI) of the prostate using a 1.5-Tesla scanner. Imaging will be interpreted by a single experienced radiologist. Only patients with lesions scored as Prostate Imaging-Reporting and Data System (PI-RADS) category 4 or 5 will be included in the study.

Participants who meet the inclusion criteria will undergo both cognitive-targeted biopsy (CTB) and magnetic resonance imaging-ultrasound fusion-targeted biopsy (FTB) during the same biopsy session. Biopsies will be performed under local or regional anesthesia using the BK3000 ultrasound system.

The study will assess predefined procedural and pathological parameters, including histopathological findings (presence or absence of malignancy and International Society of Urological Pathology [ISUP] grade group), lesion location by prostate zone and orientation, serum prostate-specific antigen and prostate-specific antigen density, lesion length, and procedure duration. Procedures will be performed by two operators (surgeon 1 and surgeon 2) according to the study protocol.

No results are reported in this section. Study outcomes will be entered in the results section after study completion.

ELIGIBILITY:
Inclusion Criteria:

Biopsy-naïve patients

Prostate-specific antigen level between 4 and 20 ng/mL

Multiparametric Magnetic Resonance Imaging Prostate Imaging-Reporting and Data System score 4 or 5

Exclusion Criteria:

Prior prostate biopsy

Prostate-specific Antigen level outside the specified range

Contraindication to Magnetic Resonance Imaging

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-28 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer Detection Rate Assessed by Histopathological Examination | During the biopsy session
  Detection of prostate cancer based on histopathological examination of biopsy core specimens obtained using cognitive-targeted biopsy and fusion-targeted biopsy. This outcome is reported as the presence or absence of prostate cancer and is not reported as a numerical score on a scale.
Clinically Significant Prostate Cancer Detection Rate Defined by International Society of Urological Pathology Grade Group | During the biopsy session
  Detection of clinically significant prostate cancer based on histopathological evaluation of biopsy specimens obtained using each biopsy technique. Clinically significant prostate cancer is defined using the International Society of Urological Pathology (ISUP) Grade Group classification, which ranges from Grade Group 1 (least aggressive) to Grade Group 5 (most aggressive). Clinically significant disease is defined as ISUP Grade Group 2 or higher. Higher ISUP grade groups indicate a worse pathological outcome.

SECONDARY OUTCOMES:
Biopsy Procedure Time Measured in Minutes | During the procedure
  Duration of each biopsy technique, measured in minutes from insertion of the ultrasound probe to completion of tissue sampling for cognitive-targeted biopsy and fusion-targeted biopsy. This outcome is a direct time measurement and not a scale-based score.
Target Lesion Length Measured on Multiparametric Magnetic Resonance Imaging | Before the biopsy procedure
  Maximum lesion length measured in millimeters on pre-biopsy multiparametric magnetic resonance imaging. This outcome is a direct physical measurement and not a score on a scale.
Procedural Metrics According to Surgeon Assignment | During the biopsy procedure
  Assessment of procedural parameters, including procedure duration, according to surgeon assignment. These outcomes are not reported as scale-based scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university hospital urology department, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No